CLINICAL TRIAL: NCT02302599
Title: Efficacy and Safety of Umbilical-cord Mesenchymal Stem Cells in Chinese Adults With Type 2 Diabetes: a Single Center, Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Mesenchymal Stem Cells to Treat Type 2 Diabetes
Acronym: UC-MSCs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yiming Mu, Director, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHIN-PLAGH-ST-003
Record Dates: First submitted 2014-11-12; First posted 2014-11-27 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes; Mesenchymal Stem Cells
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: UC-MSCs (1.5×106/kg) or the same volume of placebo (suspension liquid without UC-MSCs)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigators and participants were masked to treatment allocation. The independent data monitoring committee and the statisticians supporting the committee's activities were the only people with access to unblinded data.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Umbilical cord mesenchymal stem cells (Experimental): Patients receive Umbilical cord mesenchymal stem cells intravenous infusion for three times with an interval of 4 weeks in the absence of disease progression or unacceptable toxicity
  Interventions: Biological: Umbilical cord mesenchymal stem cells
- Controlled suspension liquid (Experimental): Patients receive Controlled suspension liquid
  Interventions: Biological: Controlled suspension liquid

INTERVENTIONS:
Biological: Umbilical cord mesenchymal stem cells — Infusion treatment
  Arms: Umbilical cord mesenchymal stem cells
Biological: Controlled suspension liquid — Infusion treatment
  Arms: Controlled suspension liquid

SUMMARY:
Umbilical cord mesenchymal stem cells indicate the therapeutic effects and safety on type 2 diabetes by characteristics of secretion and immune Immunomodulation.

DETAILED DESCRIPTION:
Umbilical cord mesenchymal stem cells can improve insulin resistance of the target tissues, reduce the islet progressive damage, ease or regenerate of the islet beta cells and improve hyperglycemic state of diabetes by secreting a variety of cytokines. It can induce damaged alpha cells differentiate into beta cells in the islet transformation to realize the islet beta cells in situ regeneration by improving microenvironment of islet beta cells. Umbilical cord mesenchymal stem cells also have immunosuppressive effect, it can promote islet cell repair and regeneration by the inhibition of T cell mediated immune response to beta cells.

ELIGIBILITY:
Inclusion Criteria:

1. 20 ≤ age ≤ 65 years;
2. Duration of type 2 diabetes ≤20 years;
3. 24.0 kg/m2 ≤ BMI ≤40.0 kg/m2;
4. Stable exogenous insulin dose between 0.5-1.0 U/Kg/Day with or without oral hypoglycemic agents (Dipeptidyl peptidase-4 (DPP-4) inhibitor, Glucagon like peptide 1 receptor (GLP-1R) agonist and Sodium-glucose co-transporter 2 (SGLT-2) inhibitor excluded) for at least 3 months;
5. 7.0% ≤ HbA1c ≤ 12.0%;
6. Fasting C-peptide ≥ 1ng/ml;
7. Willingness to participate in the trial.

Exclusion Criteria:

1. Patients with ketonuria, tumor, serum creatinine level more than 175μmol/L, myocardial infarction in the previous year, current angina or heart failure, more than one major vascular event, retinopathy requiring laser treatment, malignant hypertension, uncorrected endocrine disorder, occupations precluding insulin therapy;
2. Severe concurrent illness limiting life expectancy, inadequate understanding of the study protocol, drug abuse, pregnant willing and allergic constitution.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
The efficacy of umbilical cord mesenchymal stem cells in Chinese adults with T2D | 48 weeks from baseline
  proportion of patients with HbA1c <7.0% and daily insulin reduction ≥50% from baseline to 48 weeks

SECONDARY OUTCOMES:
Other efficacy parameter of umbilical-cord mesenchymal stem cells in Chinese adults with T2D | 48 weeks from baseline
  Changes of insulin requirement, HbA1c and proportion of patients reaching the HbA1c target (<7.0%)
Other efficacy parameter of umbilical-cord mesenchymal stem cells in Chinese adults with T2D | 48 weeks from baseline
  Change of islet β cell function and insulin resistance
safety parameter of umbilical-cord mesenchymal stem cells in Chinese adults with T2D | 48 weeks from baseline
  Fever, pruritus, nausea and vomiting, anaphylactic shock, phlebitis，tumor formation, infection, impaired liver and kidney function.

CONTACTS AND LOCATIONS:
Overall Officials: weidong HAN, Study Director — Chinese PLA General Hospital; yiming MU, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Hao H, Liu J, Shen J, Zhao Y, Liu H, Hou Q, Tong C, Ti D, Dong L, Cheng Y, Mu Y, Liu J, Fu X, Han W. Multiple intravenous infusions of bone marrow mesenchymal stem cells reverse hyperglycemia in experimental type 2 diabetes rats. Biochem Biophys Res Commun. 2013 Jul 5;436(3):418-23. doi: 10.1016/j.bbrc.2013.05.117. Epub 2013 Jun 11. PMID 23770360
- [Background] Wang XL, Lu JM, Pan CY, Mu YM, Dou JT, Ba JM. [Characteristics of the daily blood glucose profiles of impaired glucose tolerance and type 2 diabetes mellitus subjects by continuous glucose monitoring system]. Zhonghua Yi Xue Za Zhi. 2006 Mar 14;86(10):674-7. Chinese. PMID 16681924
- [Background] Si Y, Zhao Y, Hao H, Liu J, Guo Y, Mu Y, Shen J, Cheng Y, Fu X, Han W. Infusion of mesenchymal stem cells ameliorates hyperglycemia in type 2 diabetic rats: identification of a novel role in improving insulin sensitivity. Diabetes. 2012 Jun;61(6):1616-25. doi: 10.2337/db11-1141. PMID 22618776
- [Derived] Zang L, Li Y, Hao H, Liu J, Cheng Y, Li B, Yin Y, Zhang Q, Gao F, Wang H, Gu S, Li J, Lin F, Zhu Y, Tian G, Chen Y, Gu W, Du J, Chen K, Guo Q, Yang G, Pei Y, Yan W, Wang X, Meng J, Zhang S, Ba J, Lyu Z, Dou J, Han W, Mu Y. Efficacy and safety of umbilical cord-derived mesenchymal stem cells in Chinese adults with type 2 diabetes: a single-center, double-blinded, randomized, placebo-controlled phase II trial. Stem Cell Res Ther. 2022 May 3;13(1):180. doi: 10.1186/s13287-022-02848-6. PMID 35505375